CLINICAL TRIAL: NCT02881541
Title: Study of the Benefit of a Nurse (IDE) Pre and Post-operative Framework in Proctology Outpatient Surgery
Acronym: IDEPROCTO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator abandoned the project.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDEPROCTO
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Proctology; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients having Enhanced Support (Experimental): * A preoperative consultation with a nurse. This time will be dedicated to the preparation of returning home: explanation of the clinical pathway, realization of postoperative wound care, information on pain management and answer any questions the patient.
  * A nurse call on D + 1, the day after the operation to ensure the smooth running of returning home, assess postoperative pain, the correct performance of local care, answer questions from the patient, and provide advice to to limit pain .. A reminder to J2 / J3 will be produced at the request of the patient or on FDI initiative if particular difficulties are reported
  Interventions: Procedure: Enhanced support
- Patients having usual care (Experimental): no intervention will be made for this group. Patients will receive usual care respecting intern procedure
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Enhanced support
  Arms: Patients having Enhanced Support
Procedure: Usual care
  Arms: Patients having usual care

SUMMARY:
Evaluate the complement of patient care course in the development of proctology outpatient surgery (CAP) by providing:

* An additional preoperative nurse consultation day hospital
* And a phone call from a nurse at D + 1 of the operation

This corresponds to a reinforced support.

DETAILED DESCRIPTION:
Main objective of the study: help improve the care of patients in CAP including during their exit after surgery. To evaluate the quality of patient care related to this enhanced system is a lever of development assistance outpatient surgical activity.

Secondary Objectives: To evaluate the impact of this new organization

* Satisfaction of patients and caregivers
* The effectiveness of the management of patients' pain

Study period: 3 months extendable a month, no start date announced

Workforce to include 100 patients at 3 months (10 per week), 50 in the "enhanced support" group and 50 in the group "usual care"

Expected results:

The main objective evaluation criteria: Evaluation support the success rate.

Evaluation performed 45 days after the patient's surgery.

Secondary objectives: patient satisfaction (telephone questionnaire to 45 days of operation), caregivers, pain assessment (painkillers booklet completed by the patient during his first consultation), consultation or rehospitalization for emergency patients and finally degree trust the doctor vis-à-vis this new support.

ELIGIBILITY:
Inclusion Criteria:

* Patient man or woman major
* Patient primary surgery and requiring care in CAP
* Patient affiliated to a social security scheme or of such a scheme

Exclusion Criteria:

* Bedridden patient and / or not communicating
* Patient opposing his participation in the study after information
* Patient has already undergone anal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05-04 (Estimated); Primary Completion 2015-05-04 (Estimated); Study Completion 2015-05-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the success rate of the treatment using intern questionary score | Day 45 after surgery

SECONDARY OUTCOMES:
Assessment of patient satisfaction by intern phone questionary Score | Day 45 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tasseau P Angélique, MD, Principal Investigator — Fondation Hôpital Saint-Joseph

IPD SHARING:
Plan to Share IPD: Undecided